CLINICAL TRIAL: NCT06664125
Title: A Phase 2a, Multicenter, Randomized, Open-label, Active Drug-controlled Trial to Evaluate the Efficacy and Safety of JMKX003002 in End-Stage Renal Disease Patients on Hemodialysis with Hyperphosphatemia
Brief Title: Evaluate the Efficacy and Safety of JMKX003002 in End-Stage Renal Disease Patients on Hemodialysis with Hyperphosphatemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JMKX3002-H201
Record Dates: First submitted 2024-10-27; First posted 2024-10-29 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2024-10

CONDITIONS: Hyperphosphatemia
MeSH Terms: conditions — Hyperphosphatemia | interventions — Sevelamer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- JMKX003002 once daily (Experimental): JMKX003002 once daily for 4 weeks
  Interventions: Drug: JMKX003002 will be administered orally
- JMKX003002 twice daily (Experimental): JMKX003002 twice daily for 4 weeks
  Interventions: Drug: JMKX003002 will be administered orally
- Sevelamer carbonate (Active Comparator): Sevelamer carbonate three times daily for 4 weeks
  Interventions: Drug: Sevelamer carbonate

INTERVENTIONS:
Drug: JMKX003002 will be administered orally — tablets for oral administration.
  Arms: JMKX003002 once daily; JMKX003002 twice daily
Drug: Sevelamer carbonate — tablets for oral administration.
  Arms: Sevelamer carbonate

SUMMARY:
A Phase 2a, Multicenter, Randomized, Open-label, Active Drug-controlled Trial to Evaluate the Efficacy and Safety of JMKX003002 in End-Stage Renal Disease Patients on Hemodialysis with Hyperphosphatemia

DETAILED DESCRIPTION:
Evaluate the Efficacy and Safety of JMKX003002 in End-Stage Renal Disease Patients on Hemodialysis with Hyperphosphatemia

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand the procedures of this trial and provide written informed consent voluntarily;
2. Age ≥ 18 years, male or female;
3. On a stable hemodialysis regimen at a frequency of two or three times per week for at least 12 weeks prior to the screening visit;
4. Serum phosphorus within the trial-required range.

Exclusion Criteria:

1. Any history of inflammatory bowel disease or diarrheal irritable bowel syndrome;
2. Pregnant or breastfeeding;
3. Any history of a parathyroid intervention;
4. Diarrhea or loose stools occurred within 1 week prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
To preliminarily evaluate the efficacy of JMKX003002 in decreasing serum phosphorus of ESRD patients on hemodialysis | 4 weeks
  The change in serum phosphorus (sP) level from baseline to the end of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No